CLINICAL TRIAL: NCT00914771
Title: A Phase II, Randomized, Controlled, Double-blind, Multi-center, Study to Evaluate Safety and Immunogenicity of Two Doses, Administered Three Weeks Apart, of Two Monovalent H5N1 (Surface Antigen Adjuvanted With MF59C.1) Influenza Vaccines Containing 3.75 µg or 7.5 μg of H5N1 Influenza Antigen, in Non-elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Two Doses, Administered Three Weeks Apart, of Two Monovalent H5N1 Influenza Vaccines Containing 2 Doses of H5N1 Influenza Antigen, in Non-elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: V87_17
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Pandemic H5N1 Influenza
Keywords: Pandemic Influenza; H5N1; Adults and Elderly; antigen dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- H5N1 pandemic Influenza vaccine 3.75µg (Active Comparator)
  Interventions: Biological: H5N1 pandemic Influenza vaccine 3.75µg
- H5N1 pandemic Influenza vaccine 7.5µg (Active Comparator)
  Interventions: Biological: H5N1 pandemic Influenza vaccine 7.5µg

INTERVENTIONS:
Biological: H5N1 pandemic Influenza vaccine 3.75µg — 2 doses of monovalent MF59-adjuvanted H5N1 pandemic vaccine containing 3.75µg H5N1 antigen
  Arms: H5N1 pandemic Influenza vaccine 3.75µg
Biological: H5N1 pandemic Influenza vaccine 7.5µg — 2 doses of monovalent MF59-adjuvanted H5N1 pandemic vaccine containing 7.5µg H5N1 antigen
  Arms: H5N1 pandemic Influenza vaccine 7.5µg

SUMMARY:
This study aims to demonstrate the non-inferiority of two doses of H5N1 influenza antigen in non-elderly and elderly adult subjects in order to submit an extension application for a lower dose of Focetria.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 yrs of age and above on the day of enrollment.
* Individuals in good health as determined by medical history, physical examination and clinical judgment of the investigator
* Documented consent obtained after the nature of the study has been explained according to local regulatory requirements
* Individuals are able to comply with all study procedures and are available for all clinic visits scheduled in the study

Exclusion Criteria:

* Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study or who do not consent to the retention of the subject's serum samples after study completion.
* Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study
* Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Individuals who have had influenza vaccine or documented suspected influenza disease within 6 months prior to Day 1.

Laboratory-confirmed or suspected influenza disease within 6 months prior to Visit 1. "Laboratory-confirmed" includes:

1. Positive serology result
2. Positive viral culture
3. Positive rapid antigen test
4. "Suspected" influenza disease includes: subjects with influenza-like illness within the past 6 months with a household/intimate contact with "laboratory-confirmed" influenza disease

   * Individuals experiencing any acute disease or infection requiring systemic antibiotic or antiviral therapy within 6 days before vaccination (chronic antibiotic therapy for urinary tract prophylaxis is acceptable)
   * History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to influenza viral proteins, to any excipients, and to eggs (including ovalbumin), chicken protein.
   * History of any serious disease, such as:

a. Medically significant cancer (except for benign or localized skin cancer, cancer in remission for ≥10 years or localized prostate cancer that has been clinically stable for more than 2 years without treatment) b. autoimmune disease (including rheumatoid arthritis) except for Hashimoto's thyroiditis that has been clinically stable for ≥ 5 years; c. diabetes mellitus type I; d. poorly controlled diabetes mellitus type II; e. diabetes relating to genetic defects/syndromes, diseases of the exocrine pancreas, or infections; f. advanced arteriosclerotic disease; g. severe chronic obstructive pulmonary disease (COPD), i.e. GOLD stages 3 and 4; h. acute or progressive hepatic disease; i. acute or progressive renal disease; j. medically significant congestive heart failure; k. history of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (e.g., Down's syndrome)

* Known or suspected impairment/alteration of immune function, including:

  1. Receipt of immunosuppressive therapy such as oral or systemic corticosteroids, (use of inhaled, intranasal, or topical corticosteroids is allowed) or cancer chemotherapy within 60 days prior to Visit 1
  2. receipt of immunostimulants within 60 days prior to Visit 1
  3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivates within 3 months prior to Visit 1 or planned during the full length of the study
  4. HIV infection or HIV-related disease
  5. Heritable immunodeficiency
  6. Abnormalities of splenic or thymic function
* Receipt of another vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to Day 1 or planned vaccination before Day 43. Seasonal influenza vaccination is allowed 3 weeks after last study vaccination (after the blood sampling for serology on Day 43)
* Experienced body temperature ≥38.0°C (100.4°F) within 3 days prior to each study vaccination.
* Use of antipyretic/analgesic medication within 24 hours of each study vaccination
* Receipt of another investigational agent within 30 days prior to enrollment in the study or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another clinical study through the end of the study
* Pregnant or breast-feeding female
* Any positive or indeterminate pregnancy test
* If female, of childbearing potential, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry

  1. Of childbearing potential is defined as status post onset of menarche and not surgically sterile
  2. Acceptable birth control methods are defined as one or more of the following:

  i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring) ii. Barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse iii. Intrauterine device (IUD) iv. Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to the subject's study entry
* If female of childbearing potential, refusal to use an "acceptable contraceptive method" during the study including day 43.
* If female of childbearing potential, refusal to submit for pregnancy testing prior to study vaccination
* Research staff directly involved with the clinical study or family members or household members of research staff. Research staff are individuals with direct or indirect contact with study subjects, or study site personnel who have access to any study documents containing subject information. This would include receptionists, persons scheduling appointments or making screening calls, regulatory specialists, laboratory technicians, etc.
* Elective surgery or hospitalization planned during the period of study participation.
* BMI >35Kg/m2 where BMI is for obese and not for high muscle mass
* Individuals with history of substance or alcohol abuse within the past 2 years that in the opinion of the Investigator might interfere with the safety of the subject or the evaluation of the study objectives.
* Any condition, which in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Day 43 post vaccination ratio of GMTs for the 2 different vaccine groups (3.75µ / 7.5µg) including two-sided 95% confidence intervals as measured by HI and SRH in the adult and elderly population combined. | 43 days
Solicited local reactions: ecchymosis, erythema, induration, swelling and pain at injection site. | 6 weeks
Solicited systemic reactions: headache, arthralgia, chills, fatigue, malaise, myalgia, nausea, sweating and fever as measured by axillary temperature for Day 1 through 7 and Day 22 to 28 of the study. | 6 weeks

SECONDARY OUTCOMES:
Geometric mean titers/area (GMTs/GMAs) on each blood sampling days as determined by HI and SRH, and the applicable geometric mean ratios. | 6 weeks
Percentage of subjects achieving seroconversion or significant increase in antibody titer on each post-vaccination blood sampling days, as measured by HI and SRH. | 6 weeks
Percentage of subjects achieving an HI titer ≥40/ SRH area ≥25mm² on each blood sampling days. | 6 weeks
Immunogenicity, as determined by HI or SRH, will be assessed according to age-appropriate CHMP criteria (CPMP/BWP/214/96). | 6 weeks
Immunogenicity according to CBER criteria in terms of hemagglutination inhibition test in non-elderly adult and elderly subjects separately, for all post-vaccination blood sampling days and the immunogenicity according to microneutralization test | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (12):
- Poland (6):
  - NZOZ Centrum Zdrowia "Blonie", Bydgoszcz
  - Prakytka Lekarzy Rodzinnych "Salus", Katowice
  - Szpital Internistyczny, Krakow
  - Wojewodzki Specjalistyczny Szpital Dzieciecy im., Krakow
  - Samodyielny Publiczny ZOZ, Lubartów
  - NZOZ Praktyka Lekarza Rodzinnego "Eskulap", Lubin
- Turkey (Türkiye) (6):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi Ic Hastaliklan, Ankara
  - T.C.S.B. Ankara Numune Egitim ve Arastirma, Ankara
  - T.C.S.B.Ataturk Egitim ve Arastirma Hastanesi, Ankara
  - Osmangazi Universitesi Tip Fakutesi, Eskişehir
  - Enfeksiyon Hastaliklari ve Klinik Mikeoviyloji, Izmir

REFERENCES:
- [Derived] Czajka H, Unal S, Ulusoy S, Usluer G, Strus A, Sennaroglu E, Guzik J, Topeli Iskit A, Dargiewicz A, Musial D, Caylan R, Dziduch J, Eskioglu E, Hasiec B, Cwinarowiczliwa E, Belli R, Abdel-Messih IA, Beygo J, Fragapane E. A phase II, randomised clinical trial to demonstrate the non-inferiority of low-dose MF59-adjuvanted pre-pandemic A/H5N1 influenza vaccine in adult and elderly subjects. J Prev Med Hyg. 2012 Sep;53(3):136-42. PMID 23362618